CLINICAL TRIAL: NCT02754349
Title: Assessment of Pulse Wave Velocity and Augmentation Index in Patients With Atrial Fibrillation Before and After Electrical Cardioversion: a Validation Study.
Brief Title: Validation Study of Pulse Wave Velocity and Augmentation Index in Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Onze Lieve Vrouw Hospital (Other)
Responsible Party: Principal Investigator, Rogier Caluwe, Dr. Rogier Caluwé, MD, Onze Lieve Vrouw Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2014/091
Record Dates: First submitted 2016-03-28; First posted 2016-04-28 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-04

CONDITIONS: Atrial Fibrillation
Keywords: pulse wave velocity; augmentation index; central pulse pressure
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Validation (Experimental): SphygmoCor version 7, AtCor Medical, Sydney, Australia
  Interventions: Device: SphygmoCor version 7, AtCor Medical, Sydney, Australia

INTERVENTIONS:
Device: SphygmoCor version 7, AtCor Medical, Sydney, Australia — Pulse wave velocity, augmentation index and central blood pressure measurement with applanation tonometry before and after electrical cardioversion

SUMMARY:
This study aims to evaluate the reliability of measurements of arterial stiffness (pulse wave velocity (PWV), pulse wave contour analysis (PWA), central augmentation index (AIx) and pulse pressure (PP)) in atrial fibrillation (AF). For this purpose 30 AF patients scheduled for electrical cardioversion will be included. PWV and PWA measurements will be carried out before and after cardioversion.

DETAILED DESCRIPTION:
In recent years the role of arterial stiffness in the development of cardiovascular diseases has garnered attention. Indeed, arterial stiffness is now well accepted as one of the most important determinants of increasing systolic and pulse pressure thus playing a germane role in the risk of stroke and myocardial infarction. Longitudinal epidemiological studies have demonstrated the independent predictive value of arterial stiffness for cardiovascular events after adjustment for classical cardiovascular risk factors. Arterial stiffness is now a recognized intermediate endpoint for cardiovascular events. The pressure wave speed in large arteries is directly related to square root of the elastic modulus of the arterial wall (Moens-Korteweg Equation). Carotid-femoral PWV is considered the gold standard method for assessing aortic stiffness. The stiffness gradient along the aorta and central arteries, local arterial branchings and narrowing of the arterial lumen cause partial reflections of forward pressure waves traveling back to the central aorta. Forward and reflected pressure waves overlap, and the final amplitude and shape of the pulse pressure wave are determined by the phase timing of these component waves. In the aorta, forward and reflected waves are not in phase. In subjects with low PWV, reflected waves reach the central arteries during late-systole and diastole, increasing the aortic pressure in early diastole, which is physiologically advantageous. With increasing PWV, the reflected waves return earlier and impact on the central arteries during systole, thereby augmenting systolic and left ventricular pressure. This is why increasing PWV is accompanied by increasing AIx (defined as the difference between the second and first systolic pressure peak) and central PP. AIx and central PP depend on the speed of wave travel, the amplitude of reflected wave and the duration and pattern of ventricular ejection, especially with respect to change in heart rate and ventricular contractility. Where PWV is considered a direct measure of arterial stiffness, central PP and AIx are only indirect, surrogate measures. However, they provide additional information concerning wave reflections. Whether PWV, AIx and central PP measurements are influenced by the presence of AF is unknown. Studying AF patients before and after elective electrical cardioversion offers an appropriate setting to evaluate the effect of heart rate and rhytm on PWV, AIx and central PP. Patient specific confounding factors are minimized because each patient serves as its own control.

ELIGIBILITY:
Inclusion Criteria:

* man or woman, age ≥18 years
* signed written informed consent
* atrial fibrillation or flutter
* scheduled for elective electrical cardioversion

Exclusion Criteria:

* inability to understand the nature, scope and possible consequences of the study
* clinical conditions that could hamper hemodynamic measurements (absence of femoral pulse, systolic blood pressure < 90 mmHg)
* presence of prosthetic material (grafts, stents or stent-grafts) in the aorta or femoral arteries
* any condition precluding the execution of the cardioversion procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-02; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Pulse Wave Velocity (in meters per second) before and after cardioversion | immediate
  with assessment of agreement on the individual level and systematic bias using the group average before and after cardioversion

SECONDARY OUTCOMES:
Augmentation Index (in percent) before and after cardioversion | immediate
  with assessment of agreement on the individual level and systematic bias using the group average before and after cardioversion.hemodynamic parameters obtained from pulse wave analysis (including AIx en central blood pressure)
Central systolic blood pressure, diastolic blood pressure, mean arterial pressure and pulse pressure (in mmHg) before and after cardioversion and their potential effects on changes in PWV and AI after cardioversion | immediate
Heart rate (beats/min) before and after cardioversion and their potential effects on changes in PWV and AI after cardioversion. | immediate

CONTACTS AND LOCATIONS:
Locations (1):
- OLV Hospital, Aalst, Belgium

IPD SHARING:
Plan to Share IPD: No